CLINICAL TRIAL: NCT02675075
Title: DESIPHER Speech Degradation as an Indicator of Physiological Degeneration in ALS
Brief Title: DESIPHER_Speech Degradation as an Indicator of Physiological Degeneration in ALS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Florida Institute for Human and Machine Cognition (Other)
Responsible Party: Sponsor
Other Study IDs: N1902-P; I21RX001902 (NIH)
Record Dates: First submitted 2016-01-21; First posted 2016-02-05 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Voice; Voice Quality; Total Lung Capacity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans With ALS: This Cohort Study will admit all eligible, interested Veterans diagnosed with ALS who meet the inclusion criteria.

SUMMARY:
A disease called Amyotrophic lateral sclerosis (or ALS), which leads to difficulty swallowing, breathing, and movement, has been found to be higher for those serving in the military than in the general population. There are approximately 4,200 Veterans with ALS and roughly 1,000 new cases each year. When doctors attempt to determine the degree to which an ALS patient is suffering from the disease, they apply tests that are "graded" by experts. However, this approach to testing patients may not be very accurate. Researchers aim to use a system called DESIPHER to "listen" to ALS patients and find speech mistakes related to their condition. Researchers believe that, by detecting different types of errors, DESIPHER serves as a new kind of indicator of medical problems such as difficulty breathing or swallowing, without human "grading". This may also lead to a better system for automatically understanding ALS patients' speech.

DETAILED DESCRIPTION:
In 2008, Amyotrophic lateral sclerosis (ALS) or Lou Gehrig's Disease became a presumptively compensable (service connected) disease as the Institute of Medicine (IOM) Committee stated an association between the development of ALS and military service. According to the IOM report, military service increases life risk of ALS by 1.5 fold. There are approximately 4,200 Veterans with ALS and roughly 1,000 new cases each year. At the Tampa VA, since 2007, there has been a consistent rise in the number of Veterans diagnosed and treated with ALS.

Most physiological assessments that are commonly used to determine the functional status of patients with ALS require trained clinical personnel to administer and interpret the results. The investigators propose to use automatic speech understanding and machine learning software (DESIPHER) to: identify speech pathologies and use them to predict other aspects of physiological degeneration associated with ALS (e.g., respiratory difficulty or inability to swallow), and ultimately improve speech recognition for those with speech impairments. The investigators expect this to improve the ability to appropriately identify and intervene when Veterans with ALS are at risk of serious adverse medical issues such as respiratory failure and aspiration. The investigators postulate that analyzing the overall divergence of (impaired) speech, from a "normal" baseline, will prove to be more robust and a better marker for involvement than others that have been proposed.

Specific research questions to be addressed by this study are: (1) Is it possible to train a speech recognition system to adapt to increasingly more frequent language/speech errors of particular types, to produce an accurate textual transcript that would be readable by an ALS patient's caregiver or physician? (2) Are specific changes in physiological functioning: Forced Vital Capacity, tongue strength, speech velocity, weight (loss), aspiration risk, or psychological distress, reflected in different types of language/speech errors associated with ALS?

By understanding how speech functioning correlates with the degree to which other biophysical functioning has degraded, it is possible to apply a new, non-invasive measure for assessing the functionality of an ALS patient. In addition, the features associated with speech degradation it is possible to adapt existing speech recognition software to a patient's speech as it evolves over time, so that the quality of life for patients may be improved through conversation with a computer.

Respiratory failure is the main cause of morbidity and mortality in ALS patients. The investigators expect that the method of analyzing speech will present an excellent biomarker for respiratory function, as there is an expected increase in pauses during speech due to the necessity of increased frequency of respirations, a decrease in loudness, and decreased overall velocity of speech. A second major cause of death is aspiration. As the articular muscles decline, the investigators expect to note a decrease in the clarity of speech. Speech involvement often precedes swallowing involvement in ALS; thus, the investigators expect that increasing "speech divergence" will indicate potential aspiration risk.

ELIGIBILITY:
Inclusion Criteria:

* Veterans will be diagnosed with ALS
* Native speakers of U.S. English
* Will have bulbar involvement identified during initial ALS inpatient evaluation
* Forced vital capacity (FVC) of greater than 50% of the expected value for age
* An Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) Score of 40 or greater

Exclusion Criteria:

* A diagnosis of dementia
* FVC less than 50%
* Inability to speak
* Or inability to follow directions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Cohort of Veteran diagnosed with ALS seen at the Tampa VA
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel L. Phillips, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the amyotrophic lateral sclerosis (ALS) Clinic at the James A. Haley Hospital from January 2016 to November 2017
Groups:
- Healthy Controls: Anonymous Controls who were not diagnosed with any nervous system diseases.
Period: Overall Study
Arm/Group | Veterans With ALS | Healthy Controls
Started | 15 | 19
Completed | 12 | 19
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Veterans With ALS: This Cohort Study will admit all eligible, interested Veterans diagnosed with ALS who meet the inclusion criteria. Veterans were at least 18 years old, and were diagnosed with ALS, and followed at the James A Haley VA Hospital
- Healthy Controls: Healthy Controls were recruited to complete a one time vocal recording of the TIMIT and Ba repetition voice recordings.
- Total: Total of all reporting groups
Arm/Group | Veterans With ALS | Healthy Controls | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 14 | 22
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.8) | 53.3 (11.2) | 57.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 12 | 13
  Male | 14 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Tongue Strength [Mean (Standard Deviation); unit: KPa] — Population: Healthy controls were only service as baseline for Vocal recordings to minimize burden on the subjects. Tongue strength was only collected for the ALS arm.
  KPa
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 31.6 (17.2) |  | 31.6 (17.2)
Lip Strength [Mean (Standard Deviation); unit: kPa] — Population: Healthy Controls were only serving as baseline for vocal recordings. Lip strength was only collected for the ALS ARM.
  kPa
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 15.5 (9.0) |  | 15.5 (9.0)
Percent of Predicted Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Expected % Max FVC] — Population: Healthy controls only participated in vocal recording to minimize burden. This measurement was only taken for the ALS Arm of the study.
  Expected % Max FVC
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 69.1 (21.9) |  | 69.1 (21.9)
Speech Intelligence Test [Mean (Standard Deviation); unit: Percent words Intellegible] — Population: Healthy controls only participated in the Vocal recordings to minimize subject burden. This measurement was only collected for the ALS arm of the study.
  Percent words Intellegible
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 98.6 (4.5) |  | 98.6 (4.5)
ALS Functional Ratings Scale-Revised [Mean (Standard Deviation); unit: units Standardized Outcome Measu] — Standardized Outcome Measure: amyotrophic lateral sclerosis functional ratings scale-revised provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. There are 12 tasks, each task is rated from 0-4, producing a minimum score of 0 and maximum score of 48 with lower values representing a poorer outcome. Population: Healthy controls only participated in the Vocal recordings to minimize subject burden. This measurement was only collected for the ALS arm of the study.
  units Standardized Outcome Measu
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 32.5 (7.4) |  | 32.5 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Expected Lung Force Vital Capacity
Description: Forced Vital Capacity (FVC) measures the ability of the lung to move air. The change in FVC was calculated from the initial time point to either the end of study (24 months) or to final visit due to either death or loss to followup.
Time Frame: Baseline, and every 3 months up to 24 months
Population: Data for this measure were not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: % Expected Forced Vital Capacity
Arm/Group | Veterans With ALS | Healthy Controls
Number analyzed (Participants) | 9 | 0
% Expected Forced Vital Capacity | -1.25 (7.05) |

2. Secondary Outcome: Change in Tongue Strength
Description: A physiological measurement of tongue muscle strength, in multiple directions. A force measured with Iowa Oral Performance Instrument (IOPI)
Time Frame: Baseline, 3 Month intervals up to 24 months, calculated from the initial time point to either the end of study (24 months) or to final visit due to either death or loss to followup
Population: Data for this measurement was only collected on the Veterans with ALS Arm. Data for this measure were not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Veterans With ALS | Healthy Controls
Number analyzed (Participants) | 9 | 0
kPa | -.625 (5.45) |

3. Secondary Outcome: Change in Speech - as Measured by Speech Divergence
Description: A measure looking at changes in vocal characteristics away from standard language. Speech Divergence is a novel calculated measure based on identifying changes to 13 characteristics of speech. The score can range from 0-13. Zero would represent normal speech, while 13 would be distorted speech along all parameters.
Time Frame: as for outcome 2
Population: Speech Divergence is a novel calculated measure for this study based on change in vocal characteristics of 13 characteristics. Speech Divergence was not collected for the Healthy Controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Veterans With ALS
Number analyzed (Participants) | 9
score on a scale | 1.88 (1.40)

ADVERSE EVENTS:
Time Frame: Adverse Event Data was monitored from time of enrollment to end of study, loss to follow-up or death up to two years.
Groups:
- Healthy Controls: Healthy Controls were enrolled for a one time vocal recording. There was no follow-up visits for healthy controls.
Arm/Group | Veterans With ALS | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 3/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 4/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/15 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veterans With ALS (N=15) | Healthy Controls (N=19)
Tracheostomy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 — Subject was withdrawn from study after having surgery for a tracheostomy due to oxygen insufficiency.
Death due to progression of ALS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0

LIMITATIONS AND CAVEATS:
This study relied on the clinical team records to capture several variables. While there was clear protocols in place for clinicians, The ALSFRS-R and Speech Intelligibility Index both had missing data in the clinical record limiting analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT02675075/Prot_000.pdf
  • Informed Consent Form (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT02675075/ICF_001.pdf